CLINICAL TRIAL: NCT04855136
Title: An Exploratory Phase 1/2 Trial to Determine Recommended Phase 2 Dose (RP2D), Safety and Preliminary Efficacy of bb2121 (Ide-cel) Combinations in Subjects With Relapsed/Refractory Multiple Myeloma (KarMMa-7)
Brief Title: Safety and Efficacy of bb2121 (Ide-cel) Combinations in Multiple Myeloma
Acronym: KarMMa-7
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB2121-MM-007; 2020-003248-10 (EudraCT Number)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; BB2121; ide-cel; CC-220; JSMD194; BMS-986405; DPd; PVd; CAR T; KarMMa-7; Phase I; Phase II; DARA; POM; BTZ
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel; iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A- bb2121 in combination with CC-220 (± low-dose dexamethasone) (Experimental): bb2121 will be administered at a target dose of 450 x 10^6 CAR+T cells. The combination agent will be administered at different doses and/ or schedules, depending on dose limiting toxicity (DLT) evaluation.
  Interventions: Biological: BB2121; Drug: CC-220
- Arm B- bb2121 in combination with BMS-986405 (JSMD194) (Experimental): * bb2121 will be administered at a target dose of 450 x 10^6 CAR+T cells. The combination agent will be administered during Month 1 starting from the day of bb2121 infusion
  * Enrollment is closed for this Arm
  Interventions: Biological: BB2121; Drug: BMS-986405

INTERVENTIONS:
Biological: BB2121 — CAR T Cell Therapy
  Other Names: ide-cel
Drug: CC-220 — Cereblon (CRBN) E3 ligase modulatory compound (CELMoD)
  Arms: Arm A- bb2121 in combination with CC-220 (± low-dose dexamethasone)
Drug: BMS-986405 — gamma secretase inhibitor (GSI)
  Other Names: JSMD194
  Arms: Arm B- bb2121 in combination with BMS-986405 (JSMD194)

SUMMARY:
This is a global, open-label, multi-arm, multi-cohort, multi-center, phase 1/2 study to determine the safety, tolerability, efficacy, PK of bb2121 in combination with other therapies in adult subjects with R/RMM.

The following combinations will be

* Arm A will test bb2121 in combination with CC-220 (± low-dose dexamethasone)
* Arm B will test bb2121 in combination with BMS-986405 (JSMD194)

Combination agents being tested may be administered before, concurrently with and/or following (ie, maintenance) bb2121 infusion.

The study will consist of 2 parts: dose finding (Phase 1) and dose expansion (Phase 2). Dose expansion may occur in one or more arms.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

* Participant has documented diagnosis of MM and measurable disease, defined as:

  1. M-protein (serum protein electrophoresis [sPEP ≥ 0.5 g/dL] or urine protein electrophoresis [uPEP]): uPEP ≥ 200 mg/24 hours and/or
  2. Light chain MM without measurable disease in the serum or urine: Serum immunoglobulin free light chain ≥ 10 mg/dL (100 mg/L) and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Participant has received:

  1. at least 3 prior MM regimens for Arm A Cohort 1 and Arm B
  2. at least 1 but no greater than 3 prior MM regimens for Arm A Cohort 2
* Arm A Cohort 1 and Arm B: Participant has received prior treatment with an immunomodulatory agent, a proteasome inhibitor and an anti-CD38 antibody-containing regimen for at least 2 consecutive cycles.
* Arm A Cohort 2: Participant has received prior treatment with an immunomodulatory agent for at least 2 consecutive cycles.
* Evidence of PD during or within 6 months (measured from the last dose of any drug within the regimen) of completing treatment with the last antimyeloma regimen before study entry.
* Participant achieved a response (minimal response [MR] or better) to at least 1 prior treatment regimen.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

* Participant has non-secretory MM or has history of or active plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
* Participant has any of the following laboratory abnormalities:

  1. ANC and Platelets count as reported below
  2. Hemoglobin < 8 g/dL (< 4.9 mmol/L) (transfusion is not permitted within 21 days of screening)
  3. Creatinine clearance (CrCl) as reported below
  4. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
  5. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 ×upper limit of normal (ULN)
  6. Serum total bilirubin > 1.5 × ULN or > 3.0 mg/dL for participants with documented Gilbert's syndrome
  7. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) 1.5 × ULN, or history of Grade ≥ 2 hemorrhage within 30 days, or participant requires ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors)
* Participant has inadequate pulmonary function defined as oxygen saturation (SaO2) < 92% on room air.
* Participant has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) 50% of predicted normal.
* Prior exposure to CC-220 (± low-dose dexamethasone) as part of their most recent antimyeloma treatment regimen (Arm A).
* Prior exposure to BMS-986405 (JSMD194) (Arm B).
* Previous history of an allogeneic hematopoietic stem cell transplantation, treatment with any gene therapy-based therapeutic for cancer, investigational cellular therapy for cancer or BCMA targeted therapy.
* Treatment Arm A Cohort 1 and Arm B: participant has received autologous stem cell transplantation (ASCT) within 12 weeks prior to leukapheresis.
* Treatment Arm A Cohort 2: participant has received autologous stem cell transplantation (ASCT) within 12 months prior to leukapheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Does Limiting Toxicity (DLT) rates _Phase 1 | Up to 28 days from start of the combination therapy
  Percentage of participants experiencing DLTs
Complete Response Rate (CRR)_ Phase 2 | Up to 24 months
  Proportion of participants who achieved CR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed by investigator's review

SECONDARY OUTCOMES:
Incidence of Adverse Event (AEs) | Up to 24 months after the last participant received any study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Overall Response Rate (ORR) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Proportion of participants who achieved PR or better according to IMWG Uniform Response Criteria for Multiple Myeloma as assessed investigator's review
Progression-free Survival (PFS) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first study treatment (whichever is given earlier) start date to the date of either first observation of progressive disease or death due to any cause
Overall Survival (OS) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first study treatment (whichever is given earlier) start date to death due to any cause
Time to response (TTR) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first study treatment start date to the first date of documented response (PR or better)
Duration of Response (DoR) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first documentation of response (PR or better) to first documentation of PD or death due to any cause
Time to next antimyeloma treatment (TTNT) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first study treatment (whichever is given earlier) start date to first day when participant receives another antimyeloma treatment
Progression-free survival after next antimyeloma therapy (PFS2) | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time from first study treatment (whichever is given earlier) start date to documentation of PD on the next-line treatment or death from any cause, whichever is first.
Feasibility of maintenance therapy in combination with bb2121 | Up to 4 months after bb2121 infusion in the respective cohort
  Cumulative incidence of the maintenance therapy starting from bb2121 infusion with death as the competing risk
Pharmacokinetics - Cmax_Phase 1 and 2 | Up to 24 months after the last participant received any study treatment in the respective cohort
  Maximum transgene level
Pharmacokinetics - Tmax_Phase 1 and 2 | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time to maximum observed transgene level
Pharmacokinetics - AUC_Phase 1 and 2 | Up to 24 months after the last participant received any study treatment in the respective cohort
  Area under the curve of transgene level
Pharmacokinetics - AUC0-28days _Phase 1 and 2 | Up to 24 months after the last participant received any study treatment in the respective cohort
  Area under the curve of transgene level from time 0 to 28 days
Pharmacokinetics - Tlast _Phase 1 and 2 | Up to 24 months after the last participant received any study treatment in the respective cohort
  Time of last measurable transgene level

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (15):
  - Local Institution - 117, Birmingham, Alabama
  - Local Institution - 113, San Francisco, California
  - Local Institution - 101, Jacksonville, Florida
  - Local Institution - 104, Atlanta, Georgia
  - Local Institution - 120, Atlanta, Georgia
  - Local Institution - 114, Chicago, Illinois
  - Local Institution - 108, Boston, Massachusetts
  - Local Institution - 124, Boston, Massachusetts
  - Local Institution - 109, Hackensack, New Jersey
  - New York University Langone, New York, New York
  - Local Institution - 110, New York, New York
  - Local Institution - 111, Charlotte, North Carolina
  - Local Institution - 118, Philadelphia, Pennsylvania
  - Local Institution - 103, Nashville, Tennessee
  - Local Institution - 107, Houston, Texas
- Spain (2):
  - Local Institution - 201, Pamplona
  - Local Institution - 202, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com